CLINICAL TRIAL: NCT03198520
Title: REFRAME RPD Post-Market Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solvay Dental 360 (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS002
Record Dates: First submitted 2017-05-10; First posted 2017-06-26 (Actual); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Missing Teeth; Dental Wear
MeSH Terms: conditions — Anodontia; Tooth Wear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Polymer Removable Partial Denture (Other): Evaluate the change in patient Oral Health-related Quality of Life while wearing the Solvay Dental 360™ polymer Removable Partial Denture (RPD)
  Interventions: Device: Solvay Dental 360™

INTERVENTIONS:
Device: Solvay Dental 360™ — polymer Removable Partial Denture (RPD)

SUMMARY:
To evaluate the change in patient Oral Health-related Quality of Life (OHRQoL) from wearing a cobalt chrome (CoCr) removable partial denture (RPD) to wearing the Solvay Dental 360TM polymer Removable Partial Denture (RPD) for 8 weeks.

DETAILED DESCRIPTION:
Cohort study conducted in the United States & United Kingdom to assess Oral Health Related Quality of Life (OHRQoL) in patients receiving the study polymer Removable Partial Denture (RPD) as compared to their baseline Cobalt Chrome (CoCr) Removable Partial Denture (RPD) Oral Health Quality of Life (OHRQoL).

ELIGIBILITY:
Inclusion Criteria:

* with the absence of 3 or less teeth per saddle, excluding third molars
* partial denture in one arch only
* with previous denture wearing experience, and Cobalt Chrome (CoCr) Removable Partial Denture (RPD) fitted in the previous 24 months and the patient is currently and routinely wearing the denture
* With a stable oral health in terms of absence of disease activity affecting the periodontium, dental hard tissues (caries), pulp and the structural/aesthetic integrity of restored teeth
* With at least 1 posterior natural tooth occlusal stop (molar or premolar)
* Class I, Class II and Class III (Kennedy's Classification)
* Occlusal spacing (static and dynamic) around clasp assembly including the occlusal rest

Exclusion Criteria:

* Patients requiring extensive treatment prior to the provision of a removable partial denture (RPD)
* Patients with active primary disease; caries, periodontal disease or symptoms of pulpal or apical pathology to the remaining teeth
* Patients with irreversibly compromised structural/aesthetic integrity of restored teeth that cannot be restored as part of the provision of treatment.
* Patients with an opposing Removable Partial Denture (RPD). Removable Partial Denture (RPD) to only be in one arch and must oppose a full denture or a dentate arch which provides a stable occlusal relationship
* Canines are NOT to be replaced with the Removable Partial Denture's (RPDs). Patients must have their natural canines present

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Natress, DDS, Principal Investigator — Leeds School of Dentistry; Jiyeon Kim, DDS, Principal Investigator — University of Illinois Chicago
Locations (2):
- The University of Illinois Chicago College of Dentistry, Chicago, Illinois, United States
- Leeds School of Dentistry Unversity of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Solvay Dental 360™: Polymer Removable Partial Denture (RPD): Solvay Dental 360™: polymer Removable Partial Denture (RPD)
  All the participants wore Cobalt Chrome (CoCr) Removable Partial Dentures (RPD) at baseline before wearing the Solvay Dental 360™ polymer Removable Partial Denture (RPD).
Period: Overall Study
Arm/Group | Solvay Dental 360™: Polymer Removable Partial Denture (RPD)
Started | 46
Completed | 40
Not Completed | 6
Not completed — Physician Decision | 2
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 1
Not completed — Study Ended | 1

BASELINE CHARACTERISTICS:
Arm/Group | Polymer Removable Partial Denture
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.63 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 27
  More than one race | 7
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46
Education [Count of Participants; unit: Participants]
  Elementry School | 4
  High School | 17
  College | 15
  Graduate School | 8
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Oral Health-related Quality
Description: Subjects conducted the Oral Health-related Quality of Life (OHRQoL) before and after wearing the Solvay Dental 360™ polymer Removable Partial Denture (RPD). OHRQoL is a multidimensional survey which can be defined as a person's assessment of how functional, psychological, social factors, pain, or discomfort affect his/her well-being in the context of oral health. The purpose of the survey is to evaluate the change in these factors from wearing a cobalt chrome (CoCr) removable partial denture (RPD) to wearing the Solvay Dental 360™ polymer Removable Partial Denture (RPD).
  This score is calculated by a summation of the score from each question; each having the following scoring:
  Response Score Never 0 Points Hardly Ever 1 Point Occasionally 2 Points Fairly Often 3 Points Very Often 4 Points
  It ranges from 0 to 56 points. The overall scores are from the baseline Cobalt Chrome (CoCr) RPD and 8 weeks for Polymer RPD. Lower scores are better outcomes.
Time Frame: Baseline for the Cobalt Chrome (CoCr) Removable Partial Denture (RPD) and 8 weeks for Polymer Removable Partial Denture
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Solvay Dental 360™: Polymer Removable Partial Denture: Solvay Dental 360™: polymer Removable Partial Denture (RPD)
- Cobalt Chrome (CoCr) Removable Partial Denture (RPD): Cobalt Chrome (CoCr) Removable Partial Denture (RPD)
Arm/Group | Solvay Dental 360™: Polymer Removable Partial Denture | Cobalt Chrome (CoCr) Removable Partial Denture (RPD)
Number analyzed (Participants) | 40 | 44
score on a scale | 9.01 (8.14) | 14.41 (9.48)

2. Secondary Outcome: Comparison of Health of Abutment Teeth
Description: To investigate the difference in health of the abutment teeth following the use of the polymer RPD as compared to the CoCr RPD as assessed by the plaque score and gingival bleeding index.
  The plaque score is determined by assessing each tooth and the amount of plaque on the individual surfaces. The total number of plaque containing surfaces is divided by the total number of surfaces per arch of the mouth.
  Arch plaque is a subset of the whole plaque score calculated as the number of arch surfaces with plaque divided by the number of arch surfaces assessed.
  The gingival bleeding index is a designation of the degree of inflammation, as determined by a "bleeding on probing" assessment. Each tooth is probed at six sites and the bleeding is scored as present or absent. The number of sites where the bleeding is noted is divided by the total number of surfaces evaluated.
  All assessments are expressed as a percentage and an increased percentage indicates a poorer patient outcome.
Time Frame: Baseline for the Cobalt Chrome (CoCr) Removable Partial Denture (RPD) and 8 weeks for the Solvay Dental 360™: Polymer Removable Partial Denture
Measure: Mean (Standard Deviation); unit: Percentage of assessed surfaces
Arm/Group | Solvay Dental 360™: Polymer Removable Partial Denture | Cobalt Chrome (CoCr) Removable Partial Denture (RPD)
Number analyzed (Participants) | 40 | 44
Percentage of assessed surfaces
  Whole Plaque Score | 36.48 (19.95) | 39.42 (25.42)
  Arch Plaque Score | 37.39 (20.94) | 39.87 (25.10)
  Bleeding on Probing | 16.33 (15.03) | 20.40 (21.24)

3. Secondary Outcome: Operator Assessment
Description: Operator assessment of the adaptation of the polymer frame, adaption of the tissue base areas and their relationship to the frame adaptation, functional evaluation, aesthetic assessment and oral health assessment of abutment teeth and the periodontium. This assessment was done with a Likert scale at baseline for the Cobalt Chrome (CoCr) Removable Partial Denture (RPD) and visits 5, 6, 7 and 8 for the Solvay Dental 360™: Polymer Removable Partial Denture.
  This assessment of aesthetics was determined by the operator based on a five point scale rating from very dissatisfied through very satisfied. More satisfied is a better outcome.
Time Frame: Baseline for the Cobalt Chrome (CoCr) Removable Partial Denture (RPD) and visits 5 (5 weeks), 6 (6 weeks), 7 (7 weeks) and 8 (8 weeks) for the Solvay Dental 360™: Polymer Removable Partial Denture
Population: The professional (operator) is surveyed about the outcomes for the fit, function, occlusion and aesthetics.
Measure: Count of Participants; unit: Participants
Groups:
- Baseline Oral Exam: Cobalt Chrome (CoCr) Removable Partial Denture; Final Fitting: Solvay Dental 360™: Polymer Removable Partial Denture; Visit 6: Solvay Dental 360™: Polymer Removable Partial Denture; Visit 7: Solvay Dental 360™: Polymer Removable Partial Denture; Visit 8: Solvay Dental 360™: Polymer Removable Partial Denture: Operator assessment of the adaptation of the polymer frame, adaption of the tissue base areas and their relationship to the frame adaptation, functional evaluation, aesthetic assessment and oral health assessment of abutment teeth and the periodontium
Arm/Group | Baseline Oral Exam: Cobalt Chrome (CoCr) Removable Partial Denture | Final Fitting: Solvay Dental 360™: Polymer Removable Partial Denture | Visit 6: Solvay Dental 360™: Polymer Removable Partial Denture | Visit 7: Solvay Dental 360™: Polymer Removable Partial Denture | Visit 8: Solvay Dental 360™: Polymer Removable Partial Denture
Number analyzed (Participants) | 44 | 42 | 40 | 38 | 40
Participants
  Very Dissatisified | 1 | 1 | 0 | 0 | 0
  Dissatisified | 5 | 1 | 4 | 1 | 3
  Neither Satisfied or Dissatisified | 5 | 9 | 8 | 11 | 8
  Satisified | 27 | 26 | 22 | 19 | 24
  Very Satisified | 6 | 5 | 6 | 7 | 5

4. Secondary Outcome: Patient Frame Preference
Description: Patient-centered assessment of preference at the final visit for the study.
  Patients were asked to choose their preference of Removable Partial Denture based on comfort, aesthetics and chewing. Preference for a specific denture is a better outcome.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Solvay Dental 360™: Polymer Removable Partial Denture: Solvay Dental 360™ polymer Removable Partial Denture (RPD)
Arm/Group | Solvay Dental 360™: Polymer Removable Partial Denture | Cobalt Chrome (CoCr) Removable Partial Denture (RPD)
Number analyzed (Participants) | 40 | 40
Participants | 32 | 8

5. Secondary Outcome: Review for Mechanical Failure
Description: This is an evaluation of the Solvay Dental 360™ Polymer Removable Partial Denture (RPD) for chips, cracks, fractures, permanent deformation or other signs mechanical failure. The number in the reported data represents a cumulative number of Solvay Dental 360™Polymer Removable Partial Denture (RPD) devices with these mechanical failures.
  A device deficiency was defined as "the inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance."
Time Frame: Approximately 8 weeks
Population: Number of Solvay Dental 360™: Polymer Removable Partial Denture with mechanical failures
Measure: Number; unit: Number of Removable Partial Dentures
Units Other Than Participants: Polymer Removable Partial Denture
Arm/Group | Solvay Dental 360™: Polymer Removable Partial Denture
Number analyzed (Participants) | 40
Number analyzed (Polymer Removable Partial Denture) | 40
Number of Removable Partial Dentures
  Chips | 2
  Crack | 1
  Detachment | 1
  Fracture | 14
  Loss | 1
  Milling | 1

6. Secondary Outcome: Operator Assessment of Pocket Depth
Description: Oral Health parameters associated with the Removable Partial Denture (RPD) on pocket depths based on Operator assessment.
  Pocket depths are expressed in mm increments for mesial, mid, and distal locations on the lingual and buccal surfaces of the tooth. To measure pocket depth, a probe is placed beside the tooth beneath the gumline and indicates the groove between the gums and teeth. Visit 2 with the Cobalt Chrome (CoCr) Removable Partial Denture (RPD) is compared to visit 8 with the Solvay Dental 360™: Polymer Removable Partial Denture. In general, pocket depths of 1 to 3 mm indicate a healthy mouth and 4mm and greater may indicate periodontitis. The score is calculated as an average of all depths reported for all surfaces assessed.
  A lower score is a better outcome.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: pocket depths expressed in mm
Arm/Group | Solvay Dental 360™: Polymer Removable Partial Denture | Cobalt Chrome (CoCr) Removable Partial Denture (RPD)
Number analyzed (Participants) | 40 | 44
pocket depths expressed in mm | 2.19 (0.63) | 2.23 (0.64)

7. Secondary Outcome: Oral Health Parameters: Operator Assessment of Mobility:
Description: Oral Health parameters associated with the Removable Partial Denture (RPD) abutment teeth and Removable Partial Denture (RPD): mobility (measured as a categorical value of either Class I, Class II or Class III).
  Mobility of the teeth abutting the missing tooth as well as adjacent to the abutment tooth are classified via the Miller Classification as the following:
  * Class I: Tooth can be moved less than 1mm in the buccolingual or mesiodistal direction; this included no mobility
  * Class II: Tooth can be moved 1mm or more in the buccolingual or mesiodistal direction. No mobility in the occlusoapical direction (vertical mobility)
  * Class III: Tooth can be moved 1mm or more in the buccolingual or mesiodistal direction. Mobility in the occlusoapical direction is also present
  The mobility score assessment is noted as proportion of teeth that moved from a lower classification to a higher classification. Class I is a better outcome.
Time Frame: as for outcome 2
Population: Denominator is the total number of teeth assessed in the jaw that the RPD was provided for.
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Solvay Dental 360™: Polymer Removable Partial Denture | Cobalt Chrome (CoCr) Removable Partial Denture (RPD)
Number analyzed (Participants) | 40 | 44
Number analyzed (Teeth) | 219 | 233
Teeth
  Class I | 211 | 221
  Class II | 7 | 11
  Class III | 1 | 1

8. Secondary Outcome: Oral Health Parameters: Mucosal Bearing Areas
Description: Oral Health parameters associated with the Solvay Dental 360™ Removable Partial Denture (RPD): mucosal bearing areas (measured as an evaluation of bleeding on probing indicated as a categorical value of "bleeding present" or "bleeding absent", as compared to the Cobalt Chrome (CoCr) Removable Partial Denture (RPD).
  Operators were asked to rate the health of the mucosal bearing areas as poor, fair or good. The mucosal bearing area is the cushion between the denture base and the supporting bone. Good is a better outcome.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Solvay Dental 360™: Polymer Removable Partial Denture | Cobalt Chrome (CoCr) Removable Partial Denture (RPD)
Number analyzed (Participants) | 40 | 44
Participants
  Good | 36 | 40
  Fair | 4 | 4
  Poor | 0 | 0

ADVERSE EVENTS:
Time Frame: The subject will be questioned about any adverse event(s) and adverse device effect(s) at each visit up to the final 8 week visit.
Description: All adverse events, adverse device effects and or device deficiencies either observed by the Principal Investigator or reported by the subject, must be reported to the Sponsor within 24 hours. The subject will be questioned about any adverse event(s) and adverse device effect(s) at each visit up to the final 8 week visit.
Groups:
- Polymer Removable Partial Denture: Solvay Dental 360™ polymer Removable Partial Denture (RPD)
Arm/Group | Polymer Removable Partial Denture
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT03198520/Prot_000.pdf
  • Informed Consent Form (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT03198520/ICF_002.pdf
  • Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT03198520/SAP_003.pdf